CLINICAL TRIAL: NCT06436716
Title: The Second Affiliated Hospital of Nantong University, Nantong First People's Hospital, Nantong University
Brief Title: Artificial Intelligence Model for Traumatic Cervical Spinal Cord Injury Based on Radiomics and Genomics
Status: Recruiting | Type: Observational
Sponsor: Affiliated 2 Hospital of Nantong University (Other)
Responsible Party: Principal Investigator, Jiawei Jiang, Clinical Professor, Affiliated 2 Hospital of Nantong University
Other Study IDs: WuCS
Record Dates: First submitted 2024-05-15; First posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2024-05

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control, SCI-1, SCI-2, SCI-3: Control: No spinal cord injury
  Interventions: Radiation: MRI
- SCI-1: SCI-1: spinal cord injury and ASIA Grade A and B
  Interventions: Radiation: MRI
- SCI-2: SCI-2: spinal cord injury and ASIA Grade C
  Interventions: Radiation: MRI
- SCI-3: SCI-3: spinal cord injury and ASIA Grade D
  Interventions: Radiation: MRI

INTERVENTIONS:
Radiation: MRI — Every patient needs an MRI to assess spinal cord injury. This is one of the clinically necessary examinations.

SUMMARY:
Collect standardized, structured, and comprehensive disease-specific information, produce high-quality and accurate clinical data, provide a sample basis for the analysis and mining of spinal cord injury clinical big data, and establish a spinal cord injury-specific disease data platform to serve clinical work. Promote multi-center cooperation in spinal cord injury research: Establish a unified, standardized, queryable, and sharable efficient spinal cord clinical research data platform to promote multi-center cooperation in spinal cord injury clinical research and enhance the international competitiveness of this research field. Help the region to prepare for the establishment of a spinal cord injury-specific disease data platform for various hospitals in the region, forming a spinal cord injury-specific disease network center to achieve data sharing.

ELIGIBILITY:
Inclusion Criteria:

1. MRI Diagnosis of TCSCI
2. Clinic Diagnosis of TCSCI
3. The injury site must be in cervical spinal cord
4. MRI images of T2WI must be collected within 48 hours after injury
5. Complete and available imaging data, clinical data, including MRI, sex, age

Exclusion Criteria:

1. Spinal cord concussion and MRI scans have no obvious positive performance of spinal cord
2. The quality of MRI images is insufficient or there are serious motion artifacts

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: MRI image of patients within 48 hours after TCSCI in The First People's Hospital of Nantong
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2016-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
MRI image | From 2016 to 2027
  original MRI image format DICOM to Nii was based on Python (Version: 3.10.6), and those would be loaded into the MRIcroGMRI imageL software (Version: 12.2). Three spinal surgeons (with 5, 8 and 18 years of experience in interpreting spinal MRI respectively) manually depict the region of interest (ROI) of the lesion area layer by layer, to form three dimensional (3D) volume of interest (VOI). After the primary spinal surgeon finished depicting the injured spinal cord, the senior spinal surgeon checked the quality of ROI and made some adjustments.
ASIA scores | From 2016 to 2027
  ASIA scores means American Spinal Injury Association Impairment Scale. ASIA has 5 grades depends on the severity of spinal cord injury. Grade A :No sensory or motor function is preserved in sacral segments S4-S5, no sacral sparing. Grade B:Sensory but not motor function is preserved below the neurological level and includes sacral segments S4-S5, AND No motor function is preserved more than three levels below the motor level on either side of the body. Grade C: Motor function is preserved below the neurological level AND More than half of the key muscle functions below the neurological level of injury have a muscle grade of less than 3 (Grades 0-2). Grade D: Motor function is preserved below the neurological level AND At least half (half or more) of the key muscle functions below the neurological level of injury have a muscle grade ≥ 3. Grade E: If sensation and motor function are graded as normal in all segments AND the patient had prior SCI-related deficits.

SECONDARY OUTCOMES:
Age | From 2016 to 2027
  Years old, no need month nor day
Gender | From 2016 to 2027
  male and female
Weight | From 2016 to 2027
  In kilograms
Height | From 2016 to 2027
  In meters
BMI | From 2016 to 2027
  In kg/m^2

CONTACTS AND LOCATIONS:
Locations (1):
- Affiliated 2 Hospital of Nantong University, Nantong, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No